CLINICAL TRIAL: NCT05061446
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, 12-Week Dose-Ranging Study to Assess the Efficacy and Safety of Etrasimod in Japanese Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: Etrasimod Dose-Ranging Versus Placebo as Induction Therapy Study in Adult Japanese Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD334-203; C5041007 (Other: Alias Study Number)
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; APD334; Etrasimod
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Etrasimod Dose 1 (Experimental)
  Interventions: Drug: Etrasimod
- Etrasimod Dose 2 (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Etrasimod tablet by mouth, once daily for 12 weeks
  Other Names: APD334
  Arms: Etrasimod Dose 1
Drug: Etrasimod — Etrasimod tablet by mouth, once daily for 12 weeks
  Other Names: APD334
  Arms: Etrasimod Dose 2
Drug: Placebo — Etrasimod matching placebo tablet by mouth, once daily up to 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this Japan-only study is to assess the safety and efficacy of etrasimod at 2 doses in Japanese subjects with moderately to severely active ulcerative colitis (UC) when administered for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Japanese ancestry
* Diagnosed with ulcerative colitis (UC) ≥ 3 months prior to screening
* Having active UC confirmed by endoscopy
* Moderately to severely active UC

Exclusion Criteria:

* Severe extensive colitis
* Diagnosis of Crohn's disease (CD) or indeterminate colitis or the presence, history of a fistula consistent with CD
* Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (80):
- Japan (80):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kojunkai Daido Hospital, Nagoya, Aixhi-ken
  - NHO Hirosaki General Medical Center, Hirosaki-shi, Aomori
  - Hirosaki University Hospital(OCT/PFT/DLCO), Hirosaki-shi, Aomori
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Ishii Eye Clinic, Nagareyama-shi, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Ehime University Hospital, Toon-shi, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Japan Community Health Care Organization Kyushu Hospital, Kitakyushu, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Kitakyushu Municipal Medical Center, Kitakyushu-shi, Fukuoka
  - Koyanose Eye Clinic, Kitakyushu-shi, Fukuoka
  - Our Lady of the Snow St. Mary's Hospital, Kurume, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Kokura Memorial Hospital, Kutakyushu-shi, Fukuoka
  - Fukuoka Shinmizumaki Hospital, Onga-gun, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - Nakayama EYE Clinic, Fukuyama-shi, Hiroshima
  - NHO Fukuyama Medical Center, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - NHO Mito Medical Center, Higashiibaraki-gun, Ibaraki
  - Yuai Memorial Hospital, Koga-shi, Ibaraki
  - Ibaraki Seinan Medical Center Hospital, Sashima-gun, Ibaraki
  - Matsumoto Eye Clinic, Toride-shi, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura-shi, Ibaraki
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Kudo Internist Heart Clinic, Morioka, Iwate
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - JA- Kagoshima Koseiren Hospital (PET/DLCO), Kagoshima, Kagoshima-ken
  - Clinical Pathology Laboratory (Diagnostick center), Kagoshima, Kagoshima-ken
  - Sameshima Eye Clinic (OCT), Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Social Welfare Organization Imperial Gift Foundation,Inc.Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Hinaga Nishi Ophthalmology Clinic, Yokkaichi- Shi, Mie-ken
  - Mie Prefectural General Medical Center, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - JOHAS Tohoku Rosai Hospital, Sendai, Miyagi
  - Nagaoka Red Cross Hospital, Nagaoka-shi, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Medical Corporation Tokushukai Kishiwada Tokushukai Hospital, Kishiwada-shi, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Japan Community Health care Organization Osaka Hospital, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Japan Community Health care Organization Saitama Medical Center, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Hamamatsu Medical Centre, Hamamatsu, Shizuoka
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital, Hachiōji, Tokyo
  - Showa General Hospital, Kodaira-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University Hospital, Kagoshima
  - NHO Osaka National Hospital, Osaka
  - Osaka National Hospital Institutional Review Board, Osaka
  - Teikyo University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Takeuchi K, Nakase H, Hisamatsu T, Matsuoka K, Arai S, Yuasa H, Oe M, Ono R, Keating M, Gu G, Lazin K, McDonnell A, Fukuta K, Hibi T. Efficacy and safety of etrasimod in Japanese patients with ulcerative colitis: results from a phase 2 dose-ranging study. Intest Res. 2025 Apr 25. doi: 10.5217/ir.2024.00213. Online ahead of print. PMID 40275818
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 54 Japanese participants with moderate to severely active ulcerative colitis (UC) were enrolled in the study.
Groups:
- Placebo: Participants received placebo matched to etrasimod once daily, orally for 12 weeks.
- Etrasimod 1 mg: Participants received etrasimod 1 milligram (mg) tablets once daily, orally for 12 weeks.
- Etrasimod 2 mg: Participants received etrasimod 2 mg tablets once daily, orally for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Started | 18 | 17 | 19
Completed | 16 | 16 | 19
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Participant no longer available due to personal reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg | Total
Number analyzed (Participants) | 18 | 17 | 19 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (9.28) | 41.6 (14.04) | 49.5 (11.55) | 43.3 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 19
  Male | 13 | 11 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 17 | 19 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 18 | 17 | 19 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 12
Description: Clinical remission:Participants with stool frequency (SF)subscore=0(or of 1 with greater than or equal to(>=)1 point decrease from baseline,rectal bleeding(RB)subscore=0 and endoscopic score(ES)less than or equal to(<)=1(excluding friability).SF subscore:number of stools in 24-hours relative to normal number of stools for that participant in same period,score ranged from 0(normal number of stools) to 3(5 or more stools than normal),higher scores=more severity.RB subscore:most severe amount of blood passed per rectum in 24-hours,score ranged from 0(no blood seen)to 3(blood alone passes),higher scores=more severity.ES:reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy,score ranged from 0(normal or inactive disease) to 3(severe disease [spontaneous bleeding,ulceration]),higher scores=more severity.Modified Mayo score:measure disease activity for UC,score:0(normal) to 9(maximum severity),comprised subscores for SF,RB,ES.higher score=more severe disease activity.
Time Frame: Week 12
Population: FAS consisted of all randomized participants who received at least 1 dose of study treatment. Here, "number of participants analyzed" signifies only those participants who had a baseline MMS score between 5 and 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 14 | 15 | 19
Percentage of participants | 0 | 6.7 | 26.3
Statistical Analysis 1: Comparison: Placebo vs Etrasimod 1 mg; Test type: Other; Difference in percentage = 6.7, 95% CI 2-sided [-5.96 to 19.29]
Statistical Analysis 2: Comparison: Placebo vs Etrasimod 2 mg; Test type: Other; Difference in percentage = 26.3, 95% CI 2-sided [6.52 to 46.12]

2. Secondary Outcome: Percentage of Participants Who Achieved Endoscopic Improvement at Week 12
Description: Endoscopic improvement was defined as ES <= 1 (excluding friability). ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. Modified Mayo score (MMS): measure disease activity for UC, score: 0 (normal) to 9 (maximum severity),and comprised the subscores for SF, RB, ES. Higher score = more severe disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 14 | 15 | 19
Percentage of participants | 0 | 6.7 | 26.3
Statistical Analysis 1: Comparison: Placebo vs Etrasimod 1 mg; Test type: Other; Difference in percentage = 6.7, 95% CI 2-sided [-5.96 to 19.29]
Statistical Analysis 2: Comparison: Placebo vs Etrasimod 2 mg; Test type: Other; Difference in percentage = 26.3, 95% CI 2-sided [6.52 to 46.12]

3. Secondary Outcome: Percentage of Participants Who Achieved Symptomatic Remission at Week 12
Description: Symptomatic remission was defined as SF sub score = 0 (or = 1 with a >= 1 point decrease from baseline) and RB sub score = 0. SF subscore: reported number of stools in a 24-hour period relative to normal number of stools for that participant in the same period, score ranged from 0 (normal number of stools) to 3 (5 or more stools than normal), higher scores = more severity. RB subscore: reported the most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity. MMS: measure disease activity for UC, score: 0 (normal) to 9 (maximum severity), and comprised the subscores for SF, RB, ES. Higher score = more severe disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 14 | 15 | 19
Percentage of participants | 0 | 20.0 | 31.6
Statistical Analysis 1: Comparison: Placebo vs Etrasimod 1 mg; Test type: Other; Difference in percentage = 20.0, 95% CI 2-sided [-0.24 to 40.24]
Statistical Analysis 2: Comparison: Placebo vs Etrasimod 2 mg; Test type: Other; Difference in percentage = 31.6, 95% CI 2-sided [10.68 to 52.48]

4. Secondary Outcome: Percentage of Participants Who Achieved Mucosal Healing at Week 12
Description: Mucosal healing was defined as ES <= 1 (excluding friability) with histologic remission defined as a Geboes index score < 2.0). ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. The Geboes score grading system, was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicated more severe disease. Modified Mayo score (MMS): measure disease activity for UC, score: 0 (normal) to 9 (maximum severity), comprised subscores for SF, RB, ES. Higher score = more severe disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 14 | 15 | 19
Percentage of participants | 0 | 6.7 | 5.3
Statistical Analysis 1: Comparison: Placebo vs Etrasimod 1 mg; Test type: Other; Difference in percentage = 6.7, 95% CI 2-sided [-5.96 to 19.29]
Statistical Analysis 2: Comparison: Placebo vs Etrasimod 2 mg; Test type: Other; Difference in percentage = 5.3, 95% CI 2-sided [-4.78 to 15.30]

5. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response at Week 12
Description: Clinical response was defined as a >= 2-point and >= 30 percentage (%) decrease from baseline in MMS, and a >= 1-point decrease from baseline in RB subscore or an absolute RB subscore <= 1. MMS: measure disease activity for UC, score: 0 (normal) to 9 (maximum severity), and comprised the subscores for SF, RB, ES. Higher score = more severe disease activity. RB subscore: reported the most severe amount of blood passed per rectum in a 24-hour period, score ranged from 0 (no blood seen) to 3 (blood alone passes), higher scores = more severity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 14 | 15 | 19
Percentage of participants | 7.1 | 33.3 | 52.6
Statistical Analysis 1: Comparison: Placebo vs Etrasimod 1 mg; Test type: Other; Difference in percentage = 26.2, 95% CI 2-sided [-1.22 to 53.60]
Statistical Analysis 2: Comparison: Placebo vs Etrasimod 2 mg; Test type: Other; Difference in percentage = 45.5, 95% CI 2-sided [19.30 to 71.68]

6. Secondary Outcome: Percentage of Participants Who Achieved Endoscopic Normalization at Week 12
Description: Endoscopic normalization was defined as ES= 0. ES reported worst appearance of mucosa on flexible sigmoidoscopy or colonoscopy, score ranged from 0 (normal or inactive disease) to 3 (severe disease [spontaneous bleeding, ulceration]), higher scores = more severity. MMS: measure disease activity for UC, score: 0 (normal) to 9 (maximum severity), and comprised the subscores for SF, RB, ES. Higher score = more severe disease activity.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 14 | 15 | 19
Percentage of participants | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Adverse Events According to Severity
Description: An adverse event was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Severity was classified using common terminology criteria for adverse events (CTCAE), version 5.0, such as Grade 1 for mild, Grade 2 for moderate, Grade 3 for severe, Grade 4 for life-threatening, Grade 5 for death related to adverse event.
Time Frame: Day 1 of first dose of study treatment up to 4 weeks after administration of the final dose of study treatment (maximum up to 16 weeks)
Population: The safety set included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
Number analyzed (Participants) | 18 | 17 | 19
Participants
  Grade1 | 5 | 6 | 11
  Grade 2 | 5 | 3 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of first dose of study treatment up to 4 weeks after administration of the final dose of study treatment (maximum up to 16 weeks)
Arm/Group | Placebo | Etrasimod 1 mg | Etrasimod 2 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 10/18 | 9/17 | 13/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Etrasimod 1 mg (N=17) | Etrasimod 2 mg (N=19)
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Vaccination site joint pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Epiretinal membrane (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT05061446/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT05061446/SAP_001.pdf